CLINICAL TRIAL: NCT01714115
Title: Use of Eylea for the Treatment of an Optic Nerve Hemangioma
Status: No longer available | Type: Expanded Access
Sponsor: Vitreous -Retina- Macula Consultants of New York (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: Slakter 1234
Record Dates: First submitted 2012-10-16; First posted 2012-10-25 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Retinal Hemangioma
MeSH Terms: interventions — aflibercept

INTERVENTIONS:
Drug: Aflibercept — 2.0 mg Intravitreal Injection, every 2 to 4 weeks
  Other Names: Eylea, VEGF Trap-Eye

SUMMARY:
This is a single patient investigative treatment study. The patient was diagnosed with a retinal tumor in one eye. In the last 2 years, the patient has been treated with all available and conventional therapies, including intraocular injections of Avastin and Lucentis, steroids, and photodynamic therapy. Any positive results were short-term, and caused an eventual decline in central vision. Aflibercept has been shown to be effective against the growth of new vessels, secondary to macular degeneration. This study proposes that it may also be more effective in treating this particular patient and case. The study treatment plan is for 6 months initially, with the intention to continue treatment.

DETAILED DESCRIPTION:
The treatment plan will be to administer aflibercept 2.0 mg intravitreally every two to four weeks for at least six consecutive injections. Prior to initiation of therapy and at each study visit, a full ophthalmic examination, best-corrected visual acuity, and a complete review of systems to monitor for any toxicity will be performed. In addition, the investigators will perform fluorescein and indocyanine green angiography at baseline and obtain color fundus photographs as well as spectral domain OCT images to properly document the extent and degree of activity of the vascular tumor at baseline and at all study visits.

ELIGIBILITY:
Inclusion Criteria:

* retinal hemangioma
* previously treated with conventional therapies, including Avastin, Lucentis, steroid, and photodynamic therapy, with less than ideal results

Exclusion Criteria:

* ongoing reevaluation of adverse events, including inflammation, elevated intraocular pressure, or any suspected toxicity from aflibercept

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Vitreous Retina Macula Consultants of New York, New York, New York, United States

REFERENCES:
- [Background] Mennel S, Meyer CH, Callizo J. Combined intravitreal anti-vascular endothelial growth factor (Avastin) and photodynamic therapy to treat retinal juxtapapillary capillary haemangioma. Acta Ophthalmol. 2010 Aug;88(5):610-3. doi: 10.1111/j.1755-3768.2008.01449.x. Epub 2009 Feb 12. PMID 19222401
- [Background] Baba T, Kitahashi M, Kubota-Taniai M, Oshitari T, Yamamoto S. Subretinal hemorrhage after photodynamic therapy for juxtapapillary retinal capillary hemangioma. Case Rep Ophthalmol. 2011 Apr 22;2(1):134-9. doi: 10.1159/000328384. PMID 21589848